CLINICAL TRIAL: NCT01478763
Title: Analysis of Vitreous Proteins in Patients Undergoing Pars Plana Vitrectomy for Proliferative Diabetic Retinopathy
Brief Title: Vitrous Analysis in Proliferative Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Anders Kvanta (Other)
Responsible Party: Sponsor-Investigator, Anders Kvanta, Professor, St. Erik Eye Hospital
Organization: St. Erik Eye Hospital (Other)
Other Study IDs: Vitreous1
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: PDRP; vitreous; protein; vitrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vitreous samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Analysis of vitreous proteins in patients undergoing pars plana vitrectomy for proliferative diabetic retinopathy

DETAILED DESCRIPTION:
To analyse and compare vitreous proteins in patients undergoing pars plana vitrectomy for proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* proliferative diabetic retinopathy with vitreous hemorrhage

Exclusion Criteria:

* vitreous hemorrhage of other cause than proliferative diabetic retinopathy
* previous vitrectomy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing pars plana vitrectomy for proliferative diabetic retinopathy
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kvanta, PhD, Principal Investigator — St. Erik Eye Hospital
Locations (1):
- St. Erik Eye Hospital, Stockholm, NonUS, Sweden